CLINICAL TRIAL: NCT07115186
Title: Enhancing Stress Resilience and Coping Skills Among Adolescents in Rural China Through School-Based Psychological Interventions: A Cluster Randomized Controlled Trial
Brief Title: School-Based Intervention to Enhance Resilience and Stress Coping in Rural Chinese Adolescents
Acronym: EASY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: School interv. rural Adolscent
Record Dates: First submitted 2025-05-12; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Stress, Emotional; Stress-related Mental Disorders
Keywords: adolescents; randomized controlled trial; PTSD; depression; anxiety; stress-related mental disorders; rural area
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + delayed intervention (Active Comparator): Participants in this group will receive treatment as usual (TAU), which includes standard school-based support services. They will not receive the study intervention during the trial period but will be offered the full intervention after final outcome assessments. This design enables comparison between the intervention and existing standard care, while ensuring ethical access to the intervention for all participants.
  Interventions: Behavioral: wait-list condition
- intervention group (Experimental): Participants in the intervention group will receive a structured psychological program consisting of four sessions delivered over the course of one week. Each session is 40 minutes in duration and includes approximately 20 minutes of psychoeducation followed by 20 minutes of a guided writing intervention.
  The sessions will cover the following core themes: ① chronic stress and emotional regulation, ② emotional identification and acceptance, ③ cognitive emotion regulation, and ④ the cognitive triangle. Interventions will be administered by trained graduate students in clinical psychology from Peking University. These facilitators will receive specialized training on the intervention protocol, and will conduct pre-intervention assessments and participate in regular supervision. All sessions will be audio and video recorded to monitor treatment fidelity, ensure adherence to the intervention manual, and support supervision and quality assurance procedures.
  Interventions: Behavioral: Psychoeducation; Behavioral: guided written therapy

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation sessions for adolescents focus on essential topics like stress, emotional distress, and mental disorders, offering foundational knowledge to enhance their understanding and ability to manage these challenges effectively.
  Arms: intervention group
Behavioral: guided written therapy — In the guided writing intervention, students are asked to write about a recent event that triggered strong emotions on paper and, based on the requirements of each session, attempt to regulate their emotions. This approach aims to enhance students' abilities in emotional identification and emotion regulation.
  Arms: intervention group
Behavioral: wait-list condition — Participants will engage in their regular school activities, and after the intervention group completes the program, they will receive the same intervention content as the intervention group.
  Arms: TAU + delayed intervention

SUMMARY:
This study aims to evaluate the effectiveness of school-based psychological interventions in improving stress resilience and coping skills among adolescents in rural China. The intervention seeks to reduce stress-related mental health symptoms, including depression, anxiety, and post-traumatic stress, measured using validated instruments such as the Patient Health Questionnaire-9 (PHQ-9), the Generalized Anxiety Disorder 7-item scale (GAD-7), and the Child PTSD Symptom Scale for DSM-5 (CPSS-5). (See Appendix for full scale descriptions.)

Participants will be recruited from rural middle schools and randomly assigned to either an intervention group or a wait-list control group. The intervention consists of four sessions delivered over one week. Assessments will be conducted at baseline, immediately after the intervention, and again at a 3-month and 6-month follow-ups.

Researchers will use multilevel modeling (MLM) and structural equation modeling (SEM) to examine potential mediators and moderators of intervention effects, including emotion recognition, alexithymia, and coping strategies. indings are expected to provide evidence on the effectiveness and mechanisms of an existing, school-based psychological intervention tailored to the needs of adolescents in underserved rural settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled middle school students attending regular school classes
* Sufficient functional capacity in hearing, speaking, reading, and writing to participate in intervention activities and assessments.

Exclusion Criteria:

* Individuals assessed to be at high risk of suicide, based on screening or clinical judgment
* Diagnosis of severe mental disorders (e.g., psychotic disorders, severe mood disorders) that would interfere with participation or require more intensive clinical care

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 850 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD for adolescents | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The Child PTSD Symptom Scale for DSM-5 (CPSS-5) for adolescents and children (scores from 0 to 4, and total scores vary from 0 to 80). A higher score represents worse PTSD symptoms.
Depression | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The 9-item patient health questionnaire (PHQ-9) for adults (score ranges from 0 to 3, and the total score varies from 0 to 27). A higher score indicates worse depression symptoms.
Insomnia Severity | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The severity of insomnia symptoms will be assessed using the Insomnia Severity Index (ISI). This 7-item self-report measurement evaluates the severity of insomnia symptoms, the level of satisfaction with sleep, interference with daily functioning, noticeability of impairment attributed to sleep problems, and the level of distress caused by sleep disturbance (score from 0 to 4, and total score vary from 0 to 32). Each item is rated on a 5-point scale, providing a comprehensive measure of insomnia severity.
Generalized anxiety disorder | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The Generalized Anxiety Disorder-7 scale (GAD-7) for adults, adolescents, and children (scored from 0 to 3, and total score from 0 to 21). A higher score represents worse anxiety symptoms.
Alexithymia | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 22-item Peking alexithymia scale measures thoughts and behaviors that prevent people from feeling or recognizing negative emotions on a 5-point Likert scale (1 to 5, and total scores vary from 22 to 110). A higher score represents more severe alexithymia.
Emotion awareness | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 30-item Emotion awareness questionnaire measures emotion awareness on a 3-point Likert scale (1 to 3, with total scores ranging from 30 to 90). A higher score indicates better emotion awareness.

SECONDARY OUTCOMES:
Resilience | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The Connor-Davidson resilience scale is a 10-item resilience measurement scale that measures resilience on a 5-point Likert scale (scores range from 0 to 4, and the total score varies from 0 to 40). A higher score represents better resilience.
Self-esteem | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 10-item self-esteem measurement scale, Rosenberg self-esteem scale, measures self-esteem on a 4-point Likert scale (score from 0 to 3, and total score varies from 0 to 30), with higher scores indicating greater self-esteem.
Subjective Happiness Scale | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 4-item subjective happiness scale measures happiness (score from 1 to 7, and total score vary from 4 to 28). A higher score represents a happier state.
Frustration | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The 25-item frustration scale (score from 1 to 5, and total score varies from 24 to 120). A higher score represents less frustration.
Irritability | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 17-item irritability measurement scale, the Peking irritability scale, measures impulsive emotions, thoughts, and behaviors on a 5-point Likert scale (score from 1 to 5, and total score varies from 17 to 85). A higher score represents higher irritability.
Cognitive emotion regulation | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  An 18-item cognitive emotion regulation questionnaire measures the ability of emotion regulation on a 5-point Likert scale (1 to 5, and total scores vary from 18 to 90). A higher score represents more emotion regulation.
Game Addiction Scale | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 7-item game addiction scale measures game addiction on a 5-point Likert scale (score from 1 to 5, and total score varies from 7 to 35), with higher scores indicating worse game addiction.

OTHER OUTCOMES:
Suicide | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The suicidal behaviors questionnaire-revised (SBQ-R) for adolescents and children (total scores vary from 3 to 18). A higher score represents a higher suicide risk.
Subjective Units of Distress Scale | During intervention (up to 4 days)
  A single item inquires about subjective distress on a 100-point scale. A higher score represents more subjective distress.
Behavior performances | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 22-item behavior performance questionnaire measures various behavior performances such as study time, phone use, school performance, drinking alcohol, smoking, stealing, fighting, and lying.
Adverse Childhood Experiences | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 33-item adverse events questionnaire asks about adverse events before 18, including self-harm, experiencing emotional abuse, experiencing physical abuse, feeling severe distress, mental illness events (e.g., panic attack), and physical injury, etc. The score of each item ranges from 0 to 1(0=no, 1=yes), 0 to 4, or 0 to 5 (a higher score indicates a more severe adverse event)
Meaning in life | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 6-item meaning in life scale measures life meaning (score from 1 to 5, and total score varies from 6 to 30). A higher score represents a more life-meaning perception.
Non-suicidal self-injury | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The non-suicidal self-injury assessment tool (NSSI-AT-Severity) for adolescents and children (total scores vary from 5 to 16). A higher score represents a worse self-injury situation.
Somatic problems | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A somatic problems scale modified from PHQ-15, measuring various physical discomforts and pain on a 3-point Likert scale (score from 0 to 2). A higher score represents worse somatic problems.
EQ-5D-3L | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The EQ-5D-3L was developed by EuroQol to measure the health-related quality of life with 6 items. The 1~5 items are coded from 1 to 5, and the last item scores from 1 to 100. The scale will then be calculated into a value for further calculation of quality-adjusted life-years (QALYs), which will be used in the cost-effectiveness analysis.
Seeking for help | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 10-item help-seeking scale measures on a 7-point Likert scale (score from 1 to 7, and total score varies from 10 to 70), with higher scores indicating greater willingness to seek help from others.
Positive Childhood Experiences | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A questionnaire measuring positive childhood experiences with 13 items(total scores vary from 0 to 64). A higher score represents a more positive childhood experience.
Social support | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  The 12-item Multidimensional Scale of Perceived Social Support (score from 1 to 7, and total score varies from 12 to 84). A higher score represents better social support.
Adverse events during RCT | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 6-item adverse events during RCT scale measures adverse events (score from 0 to 1, and total score varies from 0 to 6). A higher score represents adverse events.
Parent-adolescent relationship | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  A 6-item parent-adolescent relationship scale measures parent-adolescent relationship (score from 0 to 4, and total score varies from 0 to 24). A higher score represents better parent-adolescent relationship.
Shame | baseline, post treatment (2 weeks after baseline), 3 month after post treatment
  An 8-item shame scale measures shame (score from 0 to 4, and total score varies from 0 to 32). A higher score represents more shame.

CONTACTS AND LOCATIONS:
Locations (1):
- Biancun middle school, Hebei, Baoding, China

IPD SHARING:
Plan to Share IPD: Undecided